CLINICAL TRIAL: NCT02098369
Title: Comparative Effectiveness of a Peer-led O2 Infoline for Patients and Caregivers (PELICAN)
Brief Title: Comparative Effectiveness of a Peer-led O2 Infoline for Patients and Caregivers
Acronym: PELICAN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: AlphaNet (Unknown); Apria Healthcare (Unknown); COPD Foundation (Other); Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other); National Jewish Health (Other); Patient-Centered Outcomes Research Institute (Other); American Association for Respiratory Care (Other)
Responsible Party: Principal Investigator, Jerry Krishnan, Professor of Medicine and Public Health; Associate Vice Chancellor for Population Health Sciences, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PCORI-CE 1304-6490
Record Dates: First submitted 2014-03-14; First posted 2014-03-28 (Estimated); Results first posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2017-11

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic obstructive pulmonary disease (COPD); Supplemental oxygen; Adherence; Telephonic education; Peer coaching
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Alkalies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Usual care (Other): Written education material (basic)
  Interventions: Behavioral: Written education material (basic)
- Proactive (Experimental): Written education material (basic) Additional education material PELICAN-Proactive [In addition to the usual care, participants will receive educational material and a proactive telephone peer coaching program (coaches call participants)]
  Interventions: Behavioral: Written education material (basic); Behavioral: Additional education material; Behavioral: PELICAN-Proactive
- Reactive (Experimental): Written education material (basic) Additional education material PELICAN-Reactive [In addition to the usual care, participants will receive educational material and a reactive telephone peer coaching program (participants call coaches)]
  Interventions: Behavioral: Written education material (basic); Behavioral: Additional education material; Behavioral: PELICAN-Reactive

INTERVENTIONS:
Behavioral: Written education material (basic) — Education material on COPD distributed to all participants.
Behavioral: Additional education material — Additional education material sent to participants in the proactive and reactive arms.
  Arms: Proactive; Reactive
Behavioral: PELICAN-Proactive — In the proactive arm, calls will be initiated by the coach. The phone calls will involve educational and social support components. PELICAN is grounded on the social cognitive theory of behavior change and seeks to improve patient adherence by addressing patient self-efficacy and outcome expectancy.
  Arms: Proactive
Behavioral: PELICAN-Reactive — Participants allocated to the reactive PELICAN group will be offered the opportunity to access the COPD Foundation Infoline toll-free.
  Arms: Reactive

SUMMARY:
About 1 million individuals in the US have a prescription for supplemental oxygen (O2). Using O2 can prolong life and increase quality of life. Patients often do not use their oxygen as prescribed, which means that they are not benefiting as much as they could be from this therapy. The purpose of this study is to evaluate whether a PEer-Led O2 Infoline for patients and CAregivers (PELICAN) will increase adherence to supplemental oxygen prescription and improve health in patients with chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
The COPD Foundation operates a peer-led telephone-based information line, but its effectiveness in promoting adherence to O2 therapy and patient-centered outcomes is unknown. Our overall hypothesis is that a patient-centered Peer-Led O2 InfoLine for patients and CAregivers (PELICAN) will increase adherence and improve health. We have developed a broad-based collaboration with patients/caregivers, advocacy groups, a national O2 supplier, and others to conduct a 3-arm pragmatic clinical trial, to evaluate the comparative effectiveness of proactive vs. reactive PELICAN interventions vs. usual care on adherence to O2 (primary outcome) and on other patient-centered outcomes (secondary outcomes).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Physician diagnosis of COPD
3. Physician prescription for home O2 for 24hrs/day, 7 days/week
4. Willing to use home O2.
5. Working telephone number.

Exclusion Criteria:

1. Unable to read and speak English.
2. Discharge to home hospice or expected survival less than 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry A Krishnan, MD, PhD, Principal Investigator — University of Illinois at Chicago
Locations (6):
- United States (6):
  - Apria Healthcare, Lake Forest, California
  - Los Angeles Biomedical Research Institute, Torrance, California
  - National Jewish Health, Denver, Colorado
  - AlphaNet, Miami, Florida
  - COPD Foundation, Miami, Florida
  - University of Illinois Hospital, Chicago, Illinois

REFERENCES:
- [Derived] Prieto-Centurion V, Holm KE, Casaburi R, Porszasz J, Basu S, Bracken NE, Gallardo R 3rd, Gonzalez V, Illendula SD, Sandhaus RA, Sullivan JL, Walsh LJ, Gerald LB, Krishnan JA. A Hybrid Effectiveness/Implementation Clinical Trial of Adherence to Long-Term Oxygen Therapy for Chronic Obstructive Pulmonary Disease. Ann Am Thorac Soc. 2023 Nov;20(11):1561-1570. doi: 10.1513/AnnalsATS.202302-104OC. PMID 37683098
- See also: Patient-Centered Outcomes Research Institute (PCORI): Funding Award details — http://www.pcori.org/research-results/2013/comparative-effectiveness-peer-led-supplemental-o2-infoline-patients-and

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care | Proactive | Reactive
Started | 142 | 154 | 148
Completed | 135 | 145 | 143
Not Completed | 7 | 9 | 5
Not completed — Withdrawal by Subject | 1 | 5 | 0
Not completed — Lost to Follow-up | 5 | 1 | 3
Not completed — Death | 1 | 1 | 1
Not completed — Other | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Proactive | Reactive | Total
Number analyzed (Participants) | 142 | 154 | 148 | 444
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.5 (9.0) | 68.0 (8.8) | 65.9 (8.4) | 66.8 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 111 | 103 | 302
  Male | 54 | 43 | 45 | 142
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 0 | 9
  Not Hispanic or Latino | 136 | 146 | 146 | 428
  Unknown or Not Reported | 2 | 3 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 2
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 25 | 31 | 26 | 82
  White | 111 | 116 | 117 | 344
  More than one race | 4 | 3 | 3 | 10
  Unknown or Not Reported | 1 | 4 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Supplemental O2 Prescription
Description: Number of individuals who used the stationary concentrator for a mean of at least 17.7 hours per day
Time Frame: 60 days
Population: All participants with evaluable data for oxygen use across all equipment.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Proactive | Reactive
Number analyzed (Participants) | 104 | 105 | 116
Participants | 77 | 73 | 97

2. Secondary Outcome: PROMIS - Physical Function
Description: Change in T-score from baseline to day 60. (A negative change in score indicates worse physical functioning.)
Time Frame: 60 days
Population: The number of participants included in the analysis for each outcome measure may not match the total number of participants enrolled in the study as some participants declined to provide responses to some outcome measures.
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Usual Care | Proactive | Reactive
Number analyzed (Participants) | 131 | 134 | 139
T-score | -0.5 (0.3) | -0.1 (0.3) | -0.2 (0.3)

3. Secondary Outcome: PROMIS - Fatigue
Description: Change in T-score from baseline to day 60. (A negative change in score indicates less fatigue.)
Time Frame: 60 days
Population: as for outcome 2
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Usual Care | Proactive | Reactive
Number analyzed (Participants) | 130 | 144 | 142
T-score | 0.1 (0.7) | -1.0 (0.6) | 0.3 (0.6)

4. Secondary Outcome: PROMIS - Emotional Distress - Anxiety
Description: Change in T-score from baseline to day 60. (A negative change in score indicates less emotional distress - anxiety.)
Time Frame: 60 days
Population: as for outcome 2
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Usual Care | Proactive | Reactive
Number analyzed (Participants) | 136 | 142 | 139
T-score | 0.3 (0.7) | -1.2 (0.7) | -0.1 (0.6)

5. Secondary Outcome: PROMIS - Sleep Disturbance
Description: Change in T-score from baseline to day 60. (A negative change in score indicates less sleep disturbance.)
Time Frame: 60 days
Population: as for outcome 2
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Usual Care | Proactive | Reactive
Number analyzed (Participants) | 135 | 142 | 140
T-score | -0.4 (0.7) | -2.1 (0.6) | -0.8 (0.7)

6. Secondary Outcome: PROMIS - Emotional Distress - Depression
Description: Change in T-score from baseline to day 60. (A negative change in score indicates less emotional distress - depression.)
Time Frame: 60 days
Population: as for outcome 2
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Usual Care | Proactive | Reactive
Number analyzed (Participants) | 135 | 141 | 141
T-score | 1.1 (0.6) | -1.8 (0.7) | 0.5 (0.7)

7. Secondary Outcome: PROMIS - Satisfaction With Social Roles and Activities
Description: Change in T-score from baseline to day 60. (A negative change in score indicates less satisfaction with social roles and activities.)
Time Frame: 60 days
Population: as for outcome 2
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Usual Care | Proactive | Reactive
Number analyzed (Participants) | 127 | 127 | 127
T-score | 0.5 (0.6) | 0.2 (0.6) | -1.2 (0.6)

8. Secondary Outcome: PROMIS - Ability to Participate in Social Roles and Activities
Description: Change in T-score from baseline to day 60. (A negative change in score indicates less ability to participate in social roles and activities.)
Time Frame: 60 days
Population: as for outcome 2
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Usual Care | Proactive | Reactive
Number analyzed (Participants) | 121 | 131 | 130
T-score | 1.0 (0.6) | 1.4 (0.6) | 0.9 (0.6)

ADVERSE EVENTS:
Arm/Group | Usual Care | Proactive | Reactive
Serious Adverse Events (participants affected / at risk) | 0/142 | 0/154 | 0/148
Other Adverse Events (participants affected / at risk) | 0/142 | 0/154 | 0/148

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes